CLINICAL TRIAL: NCT04742478
Title: ROVUS Asia Registry (Evaluate Safety and Effectiveness of Rotational Atherectomy and Intravascular Ultrasound for Heavily Calcified Coronary Lesion)
Acronym: ROVUS
Status: Recruiting | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020/2932
Record Dates: First submitted 2021-02-02; First posted 2021-02-08 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Calcification
Keywords: Atherosclerotic Calcification; Medial Artery Calcification; Rotational Atherectomy
MeSH Terms: interventions — Atherectomy, Coronary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Eligible subjects who underwent RA prior to PCI (with informed consent taken to join the study): Informed consent to be obtained either prior to PCI with rotational atherectomy planned or within 48 hours after rotational atherectomy. There will be data collection of history/demographics, laboratory results, symptoms, any serious adverse events recording for this cohort as well as a telephone follow up at 12months post rotational atherectomy.
  Interventions: Procedure: Rotational Atherectomy
- Eligible subjects who underwent RA prior to PCI (without informed consent taken to join the study): Subjects that were demised or refused to give consent will fall under this cohort. The data collection of this cohort will be done through screening of in-hospital data via available local PCI database/registry.
  Interventions: Procedure: Rotational Atherectomy

INTERVENTIONS:
Procedure: Rotational Atherectomy — Rotational atherectomy (RA) has been the most used atherectomy modality since its first inception in1988. RA uses high speed rotation (140,000 - 180,000 rpm) to ablate inelastic plaque, resulting in debris averaging 5µm in size24. The main focus of RA in the era of DES stent has been on plaque modification rather that plaque debulking with more papers showing improved PCI success rates.

SUMMARY:
Rotablation with or without other calcium debulking therapies is a safe adjunctive procedure for patients with severe coronary calcification requiring Percutaneous Coronary Intervention (PCI).

DETAILED DESCRIPTION:
This is a prospective observational multicenter cohort study of all patients with calcified coronary lesions undergoing RA in participating centres across Asia. Patients will be required to provide informed consent for data collection, including follow-up data and uploading of data on a web-based data collection platform (deidentified). Operators/ institution coordinators will fill up hardcopy or electronic (web-based) forms including patient's baseline demographics, co-morbidities, clinical data, laboratory test results, echocardiography results, coronary angiography findings with subsequent interventions performed as well as follow-up clinical and laboratory results. Note that while detailed data for individual patients will only be collected if there is informed consent, data from each institution will also be collected for aggregate data regarding procedural volume (eg. total cases with debulking therapy and specifically for ROTABLATORTM). This will give a sense of representativeness of data collected. This screening data will also include the following fields: age, gender, ethnicity, comorbidities, target vessel, prior revascularization (PCI/CABG), clinical presentation, procedural urgency, angiographic procedural details (RA and PCI) and in-hospital complication and mortality. The use of this retrospective data will require appropriate approval and will only utilize anonymized data. Only in-hospital data will be obtained and no follow up data is required from these controls. Should these data not be available in any of the participating sites, a minimum baseline demographics, procedural and inpatient outcome data with reasons for non-participation in registry should be provided for records purposes. This shall be accepted as a limitation of the study. Sub-site analysis may be performed in centres with availability of all data in this group of patients to address generalisability of the data collected.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an informed consent form
* Presence of clinical indication for percutaneous coronary intervention (PCI) and/or stent placement
* Subjects willing to comply with all research and follow-up requirements.
* Angiographic criteria (ONE of the following criteria MUST be met)

  1. Target lesions visually have at least moderate calcifications*
  2. Target lesion balloon dilatation failure
  3. Inability of devices (microcatheters, balloons or stents) to pass through the target lesion.
* Procedural criteria

  1. All patients treated with RA with or without other forms of debulking therapy

     * Moderate calcification is defined as radio-opacities noted only during cardiac cycle prior to contrast injection whereas severe calcification is defined as radio-opacities seen without cardiac motion prior to contrast injection, usually affecting both sides of the arterial lumen.

Exclusion Criteria:

* Decline to give consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with signed informed consent for percutaneous coronary intervention (PCI) and are eligible for calcium debulking treatment with rotational atherectomy with or without other forms of calcium debulking therapies will be enrolled into this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint (Procedural success) | Duration of procedure
  Procedural success defined as < 20% residual stenosis in treated segment without on-table mortality with TIMI 3 flow.

SECONDARY OUTCOMES:
Death | 1 year
  in-hospital and at 1-year follow-up
Periprocedural myocardial infarction (MI) | within 48 hours of procedure
  1. Peak CK-MB ≥ 10x ULN OR ≥ 5x ULN + new pathologic Q waves in ≥ 2 contiguous leads/ new persistent LBBB2 OR
  2. Peak Troponin T or I > 5x ULN + new pathologic Q waves/ ischemic ECG changes
Complications | within 48 hours of procedure
  Significant coronary perforation at least Type II, III or III CS based on Ellis classification
Complication | within 48 hours of procedure
  no-reflow or slow flow
Procedural time | Duration of procedure
  Time of guide engagement to removal of guide

CONTACTS AND LOCATIONS:
Overall Officials: Khung Keong Yeo, Principal Investigator — Singhealth Foundation; Shoichi Kuramitsu, Principal Investigator — Kokura Memorial Hospital
Locations (2):
- Kokura Memorial hospital, Kitakyushu, Japan
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee MS, Park KW, Shlofmitz E, Shlofmitz RA. Comparison of Rotational Atherectomy Versus Orbital Atherectomy for the Treatment of Heavily Calcified Coronary Plaques. Am J Cardiol. 2017 May 1;119(9):1320-1323. doi: 10.1016/j.amjcard.2017.01.025. Epub 2017 Feb 10. PMID 28258729
- [Background] Sharma SK, Tomey MI, Teirstein PS, Kini AS, Reitman AB, Lee AC, Genereux P, Chambers JW, Grines CL, Himmelstein SI, Thompson CA, Meredith IT, Bhave A, Moses JW. North American Expert Review of Rotational Atherectomy. Circ Cardiovasc Interv. 2019 May;12(5):e007448. doi: 10.1161/CIRCINTERVENTIONS.118.007448. PMID 31084239

DOCUMENTS (1):
  • Study Protocol (2021-01-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT04742478/Prot_000.pdf